CLINICAL TRIAL: NCT03594019
Title: Immediate Implant Placement Without Connective Tissue Graft or Socket Shield: a Randomized Controlled Clincial Trial
Brief Title: Immediate Implant Placement With Connective Tissue Graft or Socket Shield
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017_0419
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Tooth Fractures
Keywords: immediate implant placement; connective tissue graft; samll dehiscence
MeSH Terms: conditions — Tooth Fractures | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients in the control group will follow the conventional treatment protocol combined with connective tissue graft. Briefly, hopeless tooth will be extracted atraumatically. Implant will be placed in the palatal side and grafting materials will be filled in the buccal gap. Then, connective tissue graft will be harvest from palatal and fixed between bucall mocosa and bucall bone. Healing abutment will placed and collegan sponge will be used to seal the wound. After 4 months, implant impression and crown delivery will be finished.
  Interventions: Procedure: Connective tissue graft; Procedure: Immediate implant placement
- Test Group (Experimental): Patients in the test group will receive conventional immediate implant placement combined with socket shield technique. Briefly, the hopeless teeth will be splited from mesial and distal, the buccal part will be preseved and the palatal part will extracted. Implant will be placed in the palatal side and grafting materials will be filled in the buccal gap. After 4 months, implant impression and crown delivery will be finished.
  Interventions: Procedure: socket shield technique; Procedure: Immediate implant placement

INTERVENTIONS:
Procedure: Connective tissue graft — Connective tissue graft (CTG) is an oral and maxillofacial surgical procedure first described by Alan Edel in 1974. It includes the preparation the recipient site of tissue exhibiting recession by incising the gingival, obtaining the CTG from the donor site, securing the CTG at the recipient site and suturing the incised gingival tissue at both the donor and recipient sites.
  Arms: Control Group
Procedure: socket shield technique — The procedure is used to split the teeth and preserve the buccal part
  Arms: Test Group
Procedure: Immediate implant placement — The implant will be placed in the frest socket immediately after tooth extraction

SUMMARY:
The present study aims to evaluate the clinical outcomes of immediate implant placement with connective tissue graft or socket shield. Previous studies have demonstrate the intact buccal bone plate plays an important role in the stability of peri-implant soft tissue around immediately placed implants. However, it remains controverisal whether soft tissue stability could be achieved in immediate implant placement with connective tissue graft or socket shield.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of single implant treatment in anterior maxilla Patients with small dehiscence in the buccal bone plate （<2mm vertical bone loss and <5mm horizontal bone loss） Patients with natural teeth adjacent to implant site

Exclusion Criteria:

* Uncontrolled periodontal diseases Heavy smokers (>10 cigarettes/day) Unwilling to participate in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
pink esthetic score （PES） | 1 year
  An objective index introduced by Furhauser et al. 2005

SECONDARY OUTCOMES:
mucosal recession | 1 year
  the mid-buccal mucosal level change from baseline to follow-up
marginal bone loss | 1 year
  the mesial and dital marginal bone loss from baseline to follow-up evaluated by peri-apical X-ray.
pocket probing depth | 1 year
  the pocket depth at six sites around implant will be detected by periodontal probe
bleeding on probing | 1 year
  the percentage of bleeding after probing by periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China